CLINICAL TRIAL: NCT00277680
Title: A Randomized Trial Comparing Laparoscopic Bilateral Occlusion of Uterine Vessels to Uterine Fibroid Embolization for the Treatment of Symptomatic Uterine Fibroids
Brief Title: Laparoscopic Occlusion of Uterine Vessels Compared to Uterine Fibroid Embolization for Treatment of Uterine Fibroids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU22200105
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2006-01

CONDITIONS: Uterine Fibroids
Keywords: uterine fibroids; leiomyoma; laparoscopy; menorrhagia
MeSH Terms: conditions — Leiomyoma; Menorrhagia

INTERVENTIONS:
Procedure: Laparoscopic bilateral occlusion of uterine artery
Procedure: Radiological embolization (UFE)

SUMMARY:
Women with symptomatic uterine fibroids are treated either by Uterine Fibroid Embolization (UFE) or laparoscopic occlusion. The study hypothesis is that laparoscopic occlusion of uterine vessels and UFE have equal effect on bleeding symptoms. Menstrual bleeding reduction six months after treatment is the main endpoint. Secondary endpoints include participants assessment of symptom relief, and volume reduction of fibroids measured by MRI. We will also investigate possible differences in postoperative course, symptom reduction, complication, and recurrence. Patients are controlled with regular intervals up to five years after treatment.

DETAILED DESCRIPTION:
Uterine fibroid embolization (UFE)has become an alternative to hysterectomy for women with symptoms of uterine fibroids.Follow up studies of this new method have reported relief of menstrual bleeding by 85-90 % of the patients six to twelve months after treatment.Other studies have suggested laparoscopic bilateral occlusion of uterine arteries as an equal effective alternative, but to our knowledge there is no randomized studies published.

Patients recruitment : Women with symptoms of uterine fibroids referred to the clinic,who express a desire to avoid hysterectomy.

Study hypothesis: Laparoscopic occlusion of uterine vessels and UFE have equal effect on bleeding symptoms.

Gynecological examination, ultrasonography and magnetic resonance imaging (MRI) are performed preoperatively and after 1,3 and 6 months. Clinical follow up is planned after 1,3,6,12,24,36 and 60 months.A validated bleeding chard, Pictorial Blood Assessment Chart(PBAC)is filled in by the participants during the last menstruation period before treatment and before each control. A standardized questionnaire to assess the bleeding amount,pressure symptoms, pain, adverse events, other complains and patients satisfaction is also used.

ELIGIBILITY:
Inclusion Criteria:

* Menorrhagia and/or bulk symptoms associated with uterine fibroids

Exclusion Criteria:

* Malignancy
* Current or planned pregnancy
* Small submucous fibroids suitable for hysteroscopic resection
* Postmenopausal women
* Suspected or known adenomyosis
* Uterus size exceeding the umbilical level
* Contraindications against laparoscopic surgery

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2000-12; Study Completion 2010-04

PRIMARY OUTCOMES:
Reduction of menstrual bleeding six months after treatment measured by PBAC

SECONDARY OUTCOMES:
Patient assessment of symptom reduction including menorrhagia and bulk symptoms
postoperative pain
recovering time
complications
failures
recurrence
secondary interventions
Reduction in fibroids and uterus size measured by ultrasonography and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Olav Istre, MD,PhD, Study Director — Ullevål University Hospital, Dept.of Obstetrics and Gynecology; Kirsten Hald, MD, Principal Investigator — Ullevål University Hospital, Dept of Obstetrics and Gynecology; Nils-Einar Kløw, MD,PhD, Study Chair — Ullevaal University Hospital
Locations (1):
- Ullevål University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Hald K, Klow NE, Qvigstad E, Istre O. Laparoscopic occlusion compared with embolization of uterine vessels: a randomized controlled trial. Obstet Gynecol. 2007 Jan;109(1):20-7. doi: 10.1097/01.AOG.0000249602.39339.31. PMID 17197583